CLINICAL TRIAL: NCT00005213
Title: Lithium Countertransport and Blood Pressure In CARDIA and TOMHS
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1092; R01HL038256 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To conduct ancillary studies of sodium-stimulated lithium counter-transport in the Chicago components of the Coronary Heart Disease Risk Development in Young Adults (CARDIA) cohort and in the Treatment of Mild Hypertension Study (TOMHS) cohort.

DETAILED DESCRIPTION:
BACKGROUND:

CARDIA was a longitudinal study of the influence of lifestyle on coronary heart disease risk factors during the young adult and post-young-adult years, the time period during which risk for cardiovascular disease was thought to undergo crucial evolution. Four centers participated in this study. The Chicago CARDIA population consisted of 1,100 Black and white men and women age 18 to 30 at baseline, of diverse socioeconomic backgrounds.

TOMHS was a two phase double-blind randomized controlled clinical trial to determine whether pharmacologic therapy in conjunction with nutritional-hygienic intervention for persons with mild hypertension results in greater reduction of cardiovascular morbidity than nutritional-hygienic treatment alone. Four clinical centers were involved in Phase I. Participants were randomized into one of six treatment groups. Each group received nutritional-hygienic treatment plus one of the following: placebo, diuretic, alpha blocker, beta blocker, angiotensin-converting enzyme inhibitor, calcium channel blocker. Randomization was stratified to assure balance within each treatment group with regard to participants' drug treatment status prior to randomization. The primary endpoint was cardiovascular morbidity.

Abnormalities in cellular sodium metabolism have long been thought to play a role in the pathogenesis of hypertension. Techniques for measuring membrane electrolyte transport rates have been refined, providing an opportunity to characterize sodium metabolism in cells from hypertensives. The early clinical studies examined erythrocytes and leukocytes because of their easy accessibility and the possibility that they would reflect vascular tissue metabolism, and documented differences in sodium fluxes between hypertensives and normotensives. Subsequent studies have supported the early findings that abnormalities in membrane cation transport were associated with essential hypertension.

The findings up to 1988 indicated that one or more transport systems might be altered in essential hypertension but each system was not affected similarly, nor did all hypertensives show the same changes in each of the transport systems studied. The most consistent findings have been observed for sodium-stimulated lithium countertransport (LCT). Clinical and population-based studies have revealed that mean LCT is significantly elevated among hypertensives. In contrast, increased, decreased, and normal mean values have been reported for sodium cotransport, and increased or normal mean values for adenosine triphosphate (ATP)-dependent sodium-potassium pump activity.

The relationship between LCT and blood pressure has been examined in several studies. The largest of these was an epidemiological survey involving 3,800 men and women age 5 to over 75 in Gubbio, Italy. LCT was significantly and positively associated with both systolic and diastolic blood pressure in this population after controlling for age, sex, and weight, but, after controlling also for other factors known to be related to blood pressure such as serum uric acid and glucose, the relationship was inconsistently significant in this cross-sectional study. In other cross-sectional research, LCT was found to account for three percent of the variation in blood pressure in a study of healthy blood donors after adjustment for weight and age. Other cross-sectional population-based studies involving smaller numbers have shown a significant relationship between LCT and diastolic blood pressure in adolescents and in white adults, but not among Black adults; also between LCT and systolic blood pressure, but not diastolic blood pressure, in Black children and white adolescents.

Much of the data available in 1988 had been derived from small numbers in cross-sectional studies, chiefly clinical, only a few population-based. Large samples were needed to provide adequate power to detect relationships among LCT and demographic, dietary, and other factors. Prospective data were needed to assess whether LCT was an independent risk factor for future development of high blood pressure in people normotensive at baseline, whether LCT could be modified, and whether this change was associated with changes in blood pressure.

DESIGN NARRATIVE:

In the cross-sectional CARDIA investigation, studies were conducted on the relationships among lithium countertransport, blood pressure, and factors related to blood pressure such as age, sex, race, weight, body mass index, pulse, dietary factors, alcohol intake, serum glucose, triglycerides, cholesterol, high density lipoprotein cholesterol, uric acid, and ionized and total calcium. Prospective data were also collected from TOMHS to examine whether lithium countertransport was modified in mild hypertension by diet or by a combination of diet and antihypertensive drugs. Lithium countertransport was assayed in erythrocytes at the second examination in CARDIA and at baseline, 12 months, and 24 months in TOMHS.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-03; Study Completion 1990-02 (Actual)